CLINICAL TRIAL: NCT02023736
Title: Assessing Psychotherapy Outcome in Treatment as Usual Versus Treatment as Usual With the STIC Feedback System
Brief Title: Assessing Psychotherapy Outcome With Feedback
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Family Institute at Northwestern University (Other)
Collaborators: The Chicago Community Trust (Other); Jewish Child and Family Services (Unknown); Catholic Charities (Other); Community Counseling Centers of Chicago (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TFI-001
Record Dates: First submitted 2013-12-19; First posted 2013-12-30 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Individual Psychiatric Disorder; Couple Dysfunction; Family Dysfunction
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (Active Comparator): Patients in the Treatment as Usual condition receive the same psychotherapy treatment as they would were they not enrolled in the study.
  Interventions: Other: Treatment as Usual
- Treatment as Usual with the STIC (TAU + STIC) (Experimental): Patients in the TAU + STIC condition receive the treatment that they normally would from their therapist, but with the addition of the STIC measurement and feedback system.
  Interventions: Other: Systemic Therapy Inventory of Change (STIC); Other: Treatment as Usual

INTERVENTIONS:
Other: Systemic Therapy Inventory of Change (STIC) — The STIC is a computerized measurement and feedback system for use in psychotherapy. The measurement system consists of weekly questionnaires, completed on the computer, that target symptoms and functioning in a variety of domains of a clients life (e.g., individual symptoms, couple functioning, family functioning, relationship with children). The feedback system consists of a web-portal where therapists may access their clients' STIC responses, for the purposes of planning treatment, assessing progress, and discussing change with clients.
  Arms: Treatment as Usual with the STIC (TAU + STIC)
Other: Treatment as Usual — Clients receive psychotherapy treatment as planned and implemented by their psychotherapists. Exact type of treatment varies by therapist and according to client need.

SUMMARY:
This study is a comparison of client outcomes in two different types of psychotherapy treatment. In one condition clients will receive treatment-as-usual (TAU); the therapy that they would normally receive. In the other condition clients will receive treatment-as-usual but in addition their therapist will have access to empirical feedback on client progress. Clients in the feedback condition will fill out weekly online questionnaires, and their therapists will have access to a website that feeds back the results of these questionnaires. The purpose of the study is to understand the impact of providing such feedback to therapists. Participating therapists at 4 sites will offer all of their clients the opportunity to participate, and participating clients will be randomly assigned to either condition. This should result in a representative sample of client seeking treatment at these 4 Chicago-area clinics.

ELIGIBILITY:
Inclusion Criteria:

* Client seeks therapy at one of the 4 participating sites
* For Individual therapy: client must consent and complete pre-test battery before the first therapy session
* For couple therapy: both clients must consent and complete pre-test battery before the first therapy session
* For family therapy: at least one client must consent and complete pre-test battery before the first therapy session
* Clients must be 12 years of age or older
* Clients must be able to read (English or Spanish) at a 6th grade level

Exclusion Criteria:

* Clients under 12 years of age
* Clients incapable of reading at a 6th grade level
* Clients who are blind, or are have sufficiently impaired sight as to be unable to read the questions on the web portal

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Change in mental health symptoms at termination | At the termination of therapy (varies naturally case-to-case, but an average of 7 weeks) clients complete the outcome packet that asks about mental health symptoms in the previous month.
  Clients complete a self-report outcome packet measuring mental health symptoms, tailored to their demographics, including some or all of the following:
  Beck Depression Inventory II:
  Beck Anxiety Inventory:
  Outcome Questionnaire 45:
  Short-form 36 Health Survey:
  Revised Dyadic Adjustment Scale:
  Family Assessment Device:
  Strengths-Difficulties Questionnaire.

SECONDARY OUTCOMES:
Change in mental health symptoms at 6-month follow up | 6 months post termination
  Clients complete a self-report outcome packet measuring mental health symptoms, tailored to their demographics, including some or all of the following:
  Beck Depression Inventory II:
  Beck Anxiety Inventory:
  Outcome Questionnaire 45:
  Short Form 36 Health Survey:
  Revised Dyadic Adjustment Scale:
  Family Assessment Device:
  Strengths-Difficulties Questionnaire.
Change in mental health symptoms at 12-month follow-up | 12 months post termination
  Clients complete a self-report outcome packet measuring mental health symptoms, tailored to their demographics, including some or all of the following:
  Beck Depression Inventory II:
  Beck Anxiety Inventory:
  Outcome Questionnaire 45:
  Short Form 36 Health Survey:
  Revised Dyadic Adjustment Scale:
  Family Assessment Device:
  Strengths-Difficulties Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: William Pinsof, Ph.D., Principal Investigator — The Family Institute at Northwestern University
Locations (4):
- United States (4):
  - Community Counseling Centers of Chicago, Chicago, Illinois
  - Jewish Child and Family Services, Chicago, Illinois
  - Catholic Charities, Chicago, Illinois
  - The Family Institute at Northwestern University, Evanston, Illinois